CLINICAL TRIAL: NCT07183423
Title: A Pilot Double-Blind Randomized Controlled Trial on the Efficacy and Safety of a Novel Skin Barrier Product Versus Petrolatum in Individuals With Skin Barrier Dysfunction
Brief Title: Novel Skin Barrier Product Versus Petrolatum for Skin Barrier Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Makati Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Vermen Verallo-Rowell, Past Chairman of Dermatology, Current Active Consultant, Makati Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMCIRB2025-06-91
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis; Atopic Dermatitis; Xerosis; Contact Dermatitis
Keywords: Ceramides; Emollients; Skin care; Epidermis/Injuries; Coconut oil
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic; Dermatitis, Contact; Wounds and Injuries | interventions — Petrolatum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Right Arm: Applying Test Product (Experimental)
  Interventions: Other: Novel barrier repair topical product
- Left Arm: Applying no topicals (No Intervention)
- Petrolatum: Right Arm: Applying Petrolatum (Active Comparator)
  Interventions: Other: Petrolatum

INTERVENTIONS:
Other: Novel barrier repair topical product — Novel barrier product (containing ceramide, virgin coconut oil, cholesterol)
  Arms: Right Arm: Applying Test Product
Other: Petrolatum — Petrolatum application
  Arms: Petrolatum: Right Arm: Applying Petrolatum

SUMMARY:
The goal of this clinical trial is to learn if a novel barrier topical product works to treat barrier dysfunction in adults. It will also learn about the safety of the novel barrier topical product. The main questions it aims to answer are:

Does the novel barrier topical product improve skin hydration, skin sebum, redness, and pigmentation? Does it improve subjective dryness and itch? Researchers will compare the novel barrier topical product to petrolatum (a gold standard occlusive barrier repair agent) to see how they are comparable in treating skin barrier dysfunction.

Participants will:

Apply the novel barrier topical product or petrolatum twice a day for 28 days Visit the clinic once a week for checkups and tests Keep a diary of their application of the assigned product

DETAILED DESCRIPTION:
The goal of this randomized controlled trial is to determine the efficacy of a new barrier product (containing ceramide, virgin coconut oil, cholesterol) versus petrolatum in adults with skin barrier dysfunction (including mild to moderate psoriasis, atopic dermatitis, contact dermatitis, seasonal xerosis or clinically evident skin dryness).

The main questions it aims to answer are:

Primary Objective: In a pilot study, to compare the preliminary effectiveness of the test product (containing ceramides, cholesterol, coconut oil and monolaurin) versus petrolatum in improving skin barrier function, as measured by transepidermal water loss (using a Tewameter), skin hydration (using a Corneometer), skin lipids (using a Sebumeter) as well as skin erythema and pigmentation (using a Mexameter) over a four-week period.

Secondary Objectives:

To assess improvement in subjective symptoms (dryness, pruritus). To assess patient-reported outcomes, including comfort, ease of application, and overall satisfaction.

To monitor and compare any adverse events or skin reactions associated with both treatments.

Researchers will compare versus petrolatum to see if effects are comparable. Participants will upon enrollment to the study, be asked to accomplish the Personal Information Sheet and Patient Satisfaction Questionnaire. They will be taught how to mark the Visual Analogue Scale according to the degree of dryness and itch felt. They will accomplish this at Baseline, weeks 1, 2 and 4.

Non-invasive measurements will be done of: skin hydration (using Tewameter and Corneometer), skin sebum (using Sebumeter) and skin redness/pigmentation (using Mexameter) at baseline, weeks 1, 2, and 4. Pictures will also be taken of the test area at each visit.

All participants will be given a 1 or 3-week supply of either the test medication or the placebo in identical jars, color, and smell to maintain blinding. Refills will be given at each follow-up. Written instructions on how to use them will also be provided. The product will be applied twice daily on the right forearm for 28 days. The amount applied will be ⅛ teaspoon per application, with a plastic measuring spoon given for their use. They will be instructed not to apply the product to any other location. They will also be advised on the possible adverse effects and will be instructed to contact the investigator in case an adverse reaction happens. They will then be instructed to follow up after 1, 2, and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild skin barrier dysfunction, including:
* Mild to moderate atopic dermatitis, defined as SCORAD ≤ 50, and/or not currently requiring topical corticosteroids or immunomodulators.
* Mild to moderate chronic plaque psoriasis, defined as total body surface area (BSA) involved: ≤3% to 10%.
* Contact dermatitis
* Seasonal xerosis or clinically evident skin dryness
* Symmetrical or bilateral test areas available (volar forearm)
* Willing and able to provide informed consent and adhere to study procedures

Exclusion Criteria:

* Failure to meet any of the above inclusion criteria
* Severe atopic dermatitis or psoriasis requiring systemic or high-potency topical treatment
* Use of corticosteroids, calcineurin inhibitors, biologics, or phototherapy within 2 weeks
* Open wounds or evidence of secondary infection at test sites
* Pregnant or breastfeeding women
* Multiple nevi, tattoos, dense body hair in the test areas
* Debilitated or immunocompromised subjects
* Known or suspected hypersensitivity to the interventional product (or its ingredients) or petrolatum
* Refusal or failure to comply with the schedule of visits at the test site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-08-31 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Transepidermal water loss | 28 days
  using a Tewameter
Skin hydration | 28 days
  Using a Corneometer
Skin sebum | 28 days
  Using a Sebumeter
Skin erythema and pigmentation | 28 days
  Using a Mexameter

SECONDARY OUTCOMES:
Change in dryness | 28 days
  Measured by Visual Analog Scale
Change in itch | 28 days
  Measured by Visual Analog Scale
Ease in application | 28 days
  Using Patient Satisfaction Questionnaire
Skin softness and smoothness | 28 days
  Patient Satisfaction Questionnaire
Satisfaction with product | 28 days
  Using Patient Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vermen M Verallo Rowell, MD, Principal Investigator — VMV Skin Research Center & Clinics
Locations (1):
- VMV Skin Research Center & Clinics, Makati City, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in skin barrier defects and tropical barrier products. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact ccvrowell@gmail.com.